CLINICAL TRIAL: NCT00334893
Title: A Multi-Center Phase II Study of the Halichondrin B Analog E7389 in Recurrent Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer
Brief Title: Eribulin Mesylate in Treating Patients With Recurrent Ovarian Epithelial, Primary Peritoneal Cavity, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00169; NCI-2009-00169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-06027; NCI-7431; CDR0000481534; 06-027 (Other: Memorial Sloan-Kettering Cancer Center); 7431 (Other: CTEP); P30CA008748 (NIH); N01CM62206 (NIH); NCT01645592 (obsolete NCT alias); NCT01664403 (obsolete NCT alias)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — eribulin

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive eribulin mesylate IV over 15 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog

SUMMARY:
This phase II trial is studying how well eribulin mesylate works in treating patients with recurrent ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the frequency of objective response (complete and partial responses) in patients with recurrent ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer treated with E7389 (eribulin mesylate).

SECONDARY OBJECTIVES:

II. Determine the toxicity profile of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior platinum sensitivity (yes vs no).

Patients receive eribulin mesylate intravenously (IV) over 15 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer

  * Recurrent disease after ≥ 1 prior therapy, meeting 1 of the following criteria:

    * Platinum-resistant disease (progression-free interval < 6 months)
    * Platinum-sensitive disease (progression-free interval ≥ 6 months)
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mmby conventional techniques OR ≥ 10 mm by spiral CT scan
* No known brain metastasis
* Life expectancy > 2 months
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* WBC ≥ 3,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior invasive malignancy within the past 5 years except nonmelanoma skin cancer

  * Stage IA or IB endometrial cancer within the past 5 years allowed provided patient is considered disease free
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to E7389
* No HIV positivity
* No ongoing or active infection
* No cardiac arrhythmia
* No unstable angina pectoris
* No symptomatic congestive heart failure
* No psychiatric illness or social situations that would preclude study compliance
* No other uncontrolled intercurrent illness
* See Disease Characteristics
* Recovered from effects of recent surgery, radiotherapy, or chemotherapy
* No more than 2 prior cytotoxic therapies with no more than 1 non platinum, non taxane regimen
* No prior E7389
* More than 14 days since prior hormonal therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 4 weeks since prior radiotherapy
* No concurrent antitumor hormonal therapy
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No granulocyte colony-stimulating factors during the first course of study therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2006-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martee Hensley, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Hensley ML, Kravetz S, Jia X, Iasonos A, Tew W, Pereira L, Sabbatini P, Whalen C, Aghajanian CA, Zarwan C, Berlin S. Eribulin mesylate (halichondrin B analog E7389) in platinum-resistant and platinum-sensitive ovarian cancer: a 2-cohort, phase 2 study. Cancer. 2012 May 1;118(9):2403-10. doi: 10.1002/cncr.26569. Epub 2011 Sep 20. PMID 21935916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 4/17/2006 Primary Completion Date 3/13/2012 Recruitment Location at medical clinic
Groups:
- Platinum Resistant Cohort; Platinum Sensitive Cohort: Patients receive eribulin mesylate IV over 15 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  eribulin mesylate : Given IV
Period: Overall Study
Arm/Group | Platinum Resistant Cohort | Platinum Sensitive Cohort
Started | 37 | 37
Completed | 36 | 37
Not Completed | 1 | 0
Not completed — Not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Platinum-Resistant Cohort: Patients receive eribulin mesylate IV over 15 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  eribulin mesylate : Given IV
- Platinum-Sensitive Cohort: Patients receive eribulin mesylate IV over 15 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Platinum-Resistant Cohort | Platinum-Sensitive Cohort | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 26 | 48
  >=65 years | 15 | 11 | 26
Age, Continuous [Median (Full Range); unit: years] | 61 [38 to 80] | 60 [45 to 77] | 60 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Objective Response to Treatment With Eribulin Mesylate in Patients With Recurrent Ovarian, Fallopian Tube, or Peritoneal Cancer.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to a total of a year
Measure: Number; unit: participants
Groups:
- Platinum-Resistant Disease; Platinum-Sensitive Disease: Patients receive eribulin mesylate IV over 15 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  eribulin mesylate : Given IV
Arm/Group | Platinum-Resistant Disease | Platinum-Sensitive Disease
Number analyzed (Participants) | 36 | 37
participants
  Partial Response | 2 | 7
  Stable Disease | 16 | 21

2. Secondary Outcome: Toxicity Profile of Eribulin Mesylate in Patients With Recurrent Ovarian, Fallopian Tube, or Peritoneal Cancer
Description: Measured by NCI CTCAE Version 4.0. The 95% confidence intervals should be provided. Please see adverse events.
Time Frame: From the time of their first treatment with eribulin mesylate
Population: Data were not collected
Arm/Group | Platinum-Resistant Cohort | Platinum-Sensitive Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Platinum-Resistant Disease | Platinum-Sensitive Disease
Serious Adverse Events (participants affected / at risk) | 17/36 | 16/37
Other Adverse Events (participants affected / at risk) | 16/36 | 19/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum-Resistant Disease (N=36) | Platinum-Sensitive Disease (N=37)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0)
Death NOS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Death-Disease progression (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fever (Vascular disorders) | 1 (1) | 0 (0)
Hemoglobin decrease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Leukocyte count decrease/white blood cell decrease (Investigations) | 2 (2) | 3 (3)
Neutrophil count decrease (Investigations) | 10 (10) | 12 (12)
Obstruction-GI-Colon (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pain-Cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Pain-Chest wall (General disorders) | 1 (1) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 4 (4) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neurological disorder (Nervous system disorders) | 0 (0) | 1 (1)
Perforation, GI-Small Bowel NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum-Resistant Disease (N=36) | Platinum-Sensitive Disease (N=37)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Lymphocyte count decrease (Investigations) | 2 (2) | 2 (2)
Neutrophil count decrease (Investigations) | 14 (14) | 18 (18)
White blood cell decrease (Investigations) | 11 (11) | 10 (10)
AST/SGOT increase (Investigations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less